CLINICAL TRIAL: NCT00004237
Title: A Randomized Phase II Trial of Navelbine/Epirubicin Versus Navelbine/Mitozantrone Versus Cyclophosphamide/Adriamycin as Preoperative Chemotherapy in Patients With > or = 3cm Diameter Early Breast Cancer
Brief Title: Comparison of Three Combination Chemotherapy Regimens in Treating Women With Stage I or Stage II Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067481; RMNHS-TOPIC2; EU-99037
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2005-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Epirubicin; Mitoxantrone; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: mitoxantrone hydrochloride
Drug: vinorelbine tartrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying three regimens of combination chemotherapy to compare how well they work in treating women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of vinorelbine/epirubicin and vinorelbine/mitoxantrone in terms of clinical objective tumor response, clinical complete remission, and pathological complete remission in women with early stage breast cancer.
* Compare the efficacy of these 2 new regimens with an established regimen of cyclophosphamide/doxorubicin in a randomly selected control group of patients.
* Compare the toxicity and side effects of these 2 new regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to center and age (under 50 vs 50 and over). Patients are randomized to one of three treatment arms.

* Arm I: Patients receive vinorelbine IV on days 1 and 8 and epirubicin IV on day 1.
* Arm II: Patients receive vinorelbine IV on days 1 and 8 and mitoxantrone IV on day 1.
* Arm III: Patients receive doxorubicin IV and cyclophosphamide IV on day 1. Treatment continues every 3 weeks for 6 courses in the absence of unacceptable toxicity or disease progression. All patients except those who are under 50 and whose tumors are estrogen receptor negative receive oral adjuvant tamoxifen daily in addition to chemotherapy.

All patients are offered surgery following completion of chemotherapy. Radiotherapy begins within 4 weeks of completion of chemotherapy or surgery, whichever is the immediately preceding treatment.

Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 62-125 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary breast cancer that is potentially operable

  * Synchronous bilateral tumors eligible
  * At least 3 cm in maximum diameter

    * Tumors at least 2 cm eligible provided primary chemotherapy is deemed appropriate and radical surgery would otherwise be required
* No evidence of metastatic disease
* No prior breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled angina pectoris
* No heart failure
* No clinically significant uncontrolled cardiac arrhythmias
* LVEF at least 50%

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No medical or psychiatric condition that impairs ability to cope physically or psychologically with the chemotherapy regimen
* No other serious uncontrolled medical condition
* No other prior malignancy except basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-10; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian E. Smith, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - Surrey, Sutton, England, United Kingdom